CLINICAL TRIAL: NCT01178294
Title: Efficacy and Safety of B-Domain Deleted Recombinant Porcine Factor VIII (OBI-1) in the Treatment of Acquired Hemophilia A Due to Factor VIII Inhibitory Auto-antibodies
Brief Title: Study of Modified Recombinant Factor VIII (OBI-1) in Subjects With Acquired Hemophilia A
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBI-1-301
Record Dates: First submitted 2010-08-06; First posted 2010-08-10 (Estimated); Results first posted 2015-12-21 (Estimated); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Acquired Hemophilia A
Keywords: haemophilia A; blood coagulation disorders; coagulation protein disorder; hemophilia A; Acquired Hemophilia A; hematologic diseases; hemorrhagic disorders
MeSH Terms: conditions — Factor 8 deficiency, acquired; Hemophilia A; Blood Coagulation Disorders; Coagulation Protein Disorders; Hematologic Diseases; Hemorrhagic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OBI-1 (Experimental): Initial dose: 200 U/kg - additional doses at the discretion of the investigator based on FVIII activity level and clinical assessment of response to treatment (upper limit: 400 U/kg every 2 hours)
  Interventions: Biological: OBI-1

INTERVENTIONS:
Biological: OBI-1 — Intravenous infusion

SUMMARY:
This study is to test whether the study drug (OBI-1) is safe and effective for the treatment of serious bleeding episodes in people with acquired hemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from subject, trusted person or person who is legally authorized to sign on behalf of the participant (Legal Representative in U.S.), depending on local regulations
* Participants with acquired hemophilia with autoimmune inhibitory antibodies to human factor VIII with a clinical diagnosis established by the following criteria: a) Prolonged activated partial thromboplastin time (aPTT), b) Prothrombin time (PT) ≤ upper limit of normal (ULN) + 2 seconds and platelet count within normal range, c) Abnormal aPTT mixing study (patient-normal control 1:1) consistent with a factor VIII inhibitors reduced factor VIII activity level (below 10%)
* Has a serious bleeding episode, as documented by the investigator
* Be willing and able to follow all instructions and attend all study visits
* Participants taking anti-thrombotics (such as clopidogrel, heparin or heparin analogue) may be included provided three half-lives of the agent have elapsed since the last dose of the agent
* Life expectancy, prior to onset of the hemorrhagic episode, of at least 90 days
* Participants of reproductive age must use acceptable methods of contraception and if female, undergo pregnancy testing as part of the screening process

Exclusion Criteria:

* Hemodynamically unstable after blood transfusion, fluid resuscitation and pharmacologic or volume replacement pressor therapy. This hemodynamic instability is characterized by symptomatic hypotension resulting in vital organ dysfunction, such as cardiac ischemia, oliguria (urine volume <0.5 mL/kg in the previous six hours), central nervous system hypoperfusion manifested by mental status change such as confusion (unless head injury or intracranial hemorrhage is present), pulmonary compromise, and/or acidosis (manifested by pH and lactate levels)
* Has an established reason for bleeding that is not correctable
* Bleeding episode assessed likely to resolve on its own if left untreated
* Anti-OBI-1 inhibitor that exceeds 20 Bethesda Units (BU) (prospectively or retrospectively)
* Subsequent bleeding episode at the site of the initial qualifying bleeding episode within two weeks following the final OBI-1 dose for the initial qualifying bleeding episode, or subsequent bleeding episode at a different site than the initial qualifying bleeding episode within 1 week following the final OBI-1 dose for the initial qualifying bleeding episode will not be considered "new" qualifying bleeding episodes
* Prior history of bleeding disorder other than acquired hemophilia.
* Known major sensitivity to therapeutic products of pig or hamster origin; examples include therapeutics of porcine origin (e.g. previously marketed porcine factor VIII, Hyate-C®) and recombinant therapeutics prepared from hamster cells (e.g. Humira®, Advate® and Enbrel®)
* Use of hemophilia medication: rFVIIa within 3 hours prior to OBI-1 administration or aPCC treatment within 6 hours prior to OBI-1 administration
* Participation in any other clinical study within 30 days of the first OBI-1 treatment
* Anticipated need for treatment or device during the study that may interfere with the evaluation of the safety or efficacy of OBI-1, or whose safety or efficacy may be affected by OBI-1
* Is currently pregnant, breastfeeding, or planning to become pregnant or father a child during the study
* Abnormal baseline findings, any other medical condition(s) or laboratory findings that, in the opinion of the investigator, might jeopardize the subject's safety or decrease the chance of obtaining satisfactory data needed to achieve the objectives of the study
* Inability or unwillingness to comply with the study design, protocol requirements, or the follow-up procedures
* Participant of majority age under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-11-10 (Actual); Primary Completion 2013-07-01 (Actual); Study Completion 2013-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (12):
- United States (8):
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - Louisiana Center for Bleeding & Clotting Disorders, New Orleans, Louisiana
  - National Institutes of Health - Warren G. Magnuson Clinical Center, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of North Carolina at Chapel Hill Hospital, Chapel Hill, North Carolina
  - The Pennsylvania State University and Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Vanderbilt University Medical Center, Hemostasis/Hemophilia Clinic, Nashville, Tennessee
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada
- Apollo Hospitals, Chennai, Tamil Nadu, India
- United Kingdom (2):
  - Royal Free Hospital-Katharine Dormandy Haemophilia Centre and Thrombosis Unit, London, England
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, Hampshire/England

REFERENCES:
- [Result] Kruse-Jarres R, St-Louis J, Greist A, Shapiro A, Smith H, Chowdary P, Drebes A, Gomperts E, Bourgeois C, Mo M, Novack A, Farin H, Ewenstein B. Efficacy and safety of OBI-1, an antihaemophilic factor VIII (recombinant), porcine sequence, in subjects with acquired haemophilia A. Haemophilia. 2015 Mar;21(2):162-170. doi: 10.1111/hae.12627. Epub 2015 Jan 27. PMID 25623166
- [Derived] Miesbach W, Curry N, Knobl P, Percy C, Santoro R, Schmaier AH, Trautmann-Grill K, Badejo K, Chen J, Nouri M, Oberai P, Klamroth R. Real-world use of recombinant porcine sequence factor VIII in the treatment of acquired hemophilia A: EU PASS. Ther Adv Hematol. 2024 Sep 2;15:20406207241260332. doi: 10.1177/20406207241260332. eCollection 2024. PMID 39228858

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at 12 clinical sites in 4 countries (USA, Canada, UK, India). Eight sites enrolled subjects under Protocol OBI-1-301 only. Two US sites enrolled subjects under the expanded access protocol OBI-1-301a and subsequently under protocol OBI-1-301. Another 2 US sites enrolled subjects under OBI-1-301a only.
Pre-assignment Details: 29 subjects were enrolled and all were treated with OBI-1. Data from the expanded access subjects (Protocol 301a, n= 4) are included with the data from subjects enrolled under Protocol OBI-1-301 (n=25). 10 subjects discontinued prematurely and 18 completed the study. For one subject, the completion status could not be verified.
Period: Overall Study
Arm/Group | OBI-1
Started | 29 (25 subjects enrolled under OBI-1-301 + 4 subjects enrolled under expanded access OBI-1-301a.)
Completed | 18
Not Completed | 11
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 2
Not completed — Lack of Efficacy | 1
Not completed — Death | 1
Not completed — Development of inhibitors to OBI-1 | 1
Not completed — Subject status is terminal | 1
Not completed — Completion status could not be verified | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population comprises all 29 treated subjects (=safety analysis set).
Arm/Group | OBI-1
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (13.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 19
Region of Enrollment [Count of Participants; unit: Participants] — Of 16 subjects enrolled in the US, 12 were enrolled under Protocol 301 and 4 were enrolled under the expanded access Protocol 301a.
  Participants
    United States | 16
    Canada | 5
    United Kingdom | 4
    India | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Serious Bleeding Episodes Responsive to OBI-1
Description: The initial serious ("qualifying") bleeding episode for each subject was analyzed for the primary efficacy outcome measure. A 'positive response' is defined as 'effective' (bleeding stopped with clinical control and FVIII levels of 50% or higher ) or 'partially effective' (bleeding reduced with clinical stabilization and FVIII levels of 20% or higher) control of bleeding, as determined by the investigator using a 4-point rating scale (effective - partially effective - poorly effective - not effective). 'Poorly effective' is defined as 'bleeding slightly reduced or unchanged and FVIII levels of less than 50%'. 'Not effective' is defined as 'bleeding worsening and FVIII levels of less than 50%'.
Time Frame: 24 hours after initiation of treatment
Population: Intent to Treat (ITT) population = 29 subjects with initial serious bleeding episodes
Measure: Number (95% Confidence Interval); unit: percentage of serious bleeding episodes
Units Other Than Participants: Initial Serious Bleeding Episodes
Arm/Group | OBI-1
Number analyzed (Participants) | 29
Number analyzed (Initial Serious Bleeding Episodes) | 29
percentage of serious bleeding episodes | 100 [88.1 to 100]
Statistical Analysis 1: Comparison: OBI-1; Summary statistics for the percentage of participants with serious bleeding episodes responsive at 24 hours after the initiation of treatment are presented, along with the 95% confidence interval (two-sided 95% Clopper-Pearson confidence interval); Test type: Superiority or Other; p < 0.001, one-sided binomial exact test

2. Secondary Outcome: Overall Percentage of Serious Bleeding Episodes Successfully Controlled With OBI-1 Therapy, as Assessed by the Investigator
Description: Treatment success was defined as control of qualifying bleeding episode at the time of final treatment dosing. A serious bleeding episode was considered 'successfully controlled' if the investigator had checked 'completed OBI-1 therapy as treatment success' on the eCRF.
Time Frame: At the time of final treatment dosing (varied from participant to participant depending on bleeding episodes)
Population: ITT population = 29 subjects with initial serious bleeding episodes (BEs)
Measure: Number (95% Confidence Interval); unit: percentage of serious bleeding episodes
Units Other Than Participants: Initial Serious Bleeding Episodes
Arm/Group | OBI-1
Number analyzed (Participants) | 29
Number analyzed (Initial Serious Bleeding Episodes) | 29
percentage of serious bleeding episodes | 86.2 [68.3 to 96.1]

3. Secondary Outcome: Percentage of Serious Bleeding Episodes Responsive to OBI-1 Therapy at Designated Assessment Time Points After the Initiation of Therapy, as Assessed by the Investigator
Description: A 'positive response' is defined as 'effective' (bleeding stopped with clinical control and FVIII levels of 50% or higher ) or 'partially effective' (bleeding reduced with clinical stabilization and FVIII levels of 20% or higher) control of bleeding, as determined by the investigator using a 4-point rating scale (effective - partially effective - poorly effective - not effective). 'Poorly effective' is defined as 'bleeding slightly reduced or unchanged and FVIII levels of less than 50%'. 'Not effective' is defined as 'bleeding worsening and FVIII levels of less than 50%'.
Time Frame: 8 hours
Population: 21 subjects of the ITT population (n=29) had responses available at 8 hours after initial infusion of OBI-1.
Measure: Number (95% Confidence Interval); unit: percentage of serious bleeding episodes
Units Other Than Participants: Responses Available at 8 hrs
Arm/Group | OBI-1
Number analyzed (Participants) | 21
Number analyzed (Responses Available at 8 hrs) | 21
percentage of serious bleeding episodes | 95.2 [76.2 to 99.9]

4. Secondary Outcome: Percentage of Serious Bleeding Episodes Responsive to OBI-1 Therapy at Designated Assessment Time Points After the Initiation of Therapy, as Assessed by the Investigator
Description: as for outcome 3
Time Frame: 16 hours
Population: 19 subjects of the ITT population (n=29) had responses available at 16 hours after initial infusion of OBI-1.
Measure: Number (95% Confidence Interval); unit: percentage of serious bleeding episodes
Units Other Than Participants: Responses Available at 16 hrs
Arm/Group | OBI-1
Number analyzed (Participants) | 19
Number analyzed (Responses Available at 16 hrs) | 19
percentage of serious bleeding episodes | 100 [82.4 to 100]

5. Secondary Outcome: Frequency of Infusions of OBI-1 Required to Successfully Control Qualifying Bleeding Episodes
Description: 'Frequency of infusions' was calculated as the 'average number of infusions per day'. 'Qualifying bleeding episode' was defined as the 'initial, serious bleeding episode'.
Time Frame: Time of successful control of qualifying bleeding episode (varied from participant to participant)
Population: The analysis was performed in 25 of 29 participants in the ITT population whose 'qualifying' bleeding episode was controlled successfully.
Measure: Mean (Standard Deviation); unit: average number of infusions per day
Arm/Group | OBI-1
Number analyzed (Participants) | 25
average number of infusions per day | 2.10 (1.109)

6. Secondary Outcome: Total Dose of OBI-1 Required to Successfully Control 'Qualifying' Bleeding Episodes
Description: 'Qualifying bleeding episode' was defined as the 'initial, serious bleeding episode'.
Time Frame: Time of successful control of qualifying bleeding episode (varied from participant to participant)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: dose in U/kg
Arm/Group | OBI-1
Number analyzed (Participants) | 25
dose in U/kg | 2683.2 (2928.61)

7. Secondary Outcome: Total Number of Infusions of OBI-1 Required to Successfully Control 'Qualifying' Bleeding Episodes
Description: 'Qualifying bleeding episode' was defined as the 'initial, serious bleeding episode'. A serious bleeding episode was considered 'successfully controlled' if the investigator had checked 'completed OBI-1 therapy as treatment success' on the eCRF.
Time Frame: Time of successful control of qualifying bleeding episode (varied from participant to participant)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: infusions per participant
Arm/Group | OBI-1
Number analyzed (Participants) | 25
infusions per participant | 15.4 (12.64)

8. Secondary Outcome: Correlation Between Positive Response to OBI-1 Therapy at 8 Hours and Eventual Control of Serious Bleeding Episodes at 24 Hours
Time Frame: 24 hours
Population: Of 21 subjects in the ITT population (n=29) with responses available at 8 hours after initial infusion of OBI-1, 20 had a positive response.
Measure: Number; unit: subjects with eventual bleed control
Arm/Group | OBI-1
Number analyzed (Participants) | 21
subjects with eventual bleed control | 17

9. Secondary Outcome: Correlation Between Response to OBI-1 Therapy at 16 Hours and Eventual Control of Serious Bleeding Episodes at 24 Hours
Time Frame: 24 hours
Population: All 19 subjects in the ITT population (n=29) who had responses available at 16 hours after initial infusion of OBI-1 had a positive response.
Measure: Number; unit: subjects with eventual bleed control
Arm/Group | OBI-1
Number analyzed (Participants) | 19
subjects with eventual bleed control | 17

10. Secondary Outcome: Correlation Between Response to OBI-1 Therapy at Specified Time Points and Eventual Control of Serious Bleeding Episodes at 24 Hours
Time Frame: 24 hours
Population: 29 subjects (ITT population) had responses available at 24 hours after initial infusion of OBI-1.
Measure: Number; unit: participants with bleeds controlled
Arm/Group | OBI-1
Number analyzed (Participants) | 29
participants with bleeds controlled | 25

11. Secondary Outcome: Correlation Between the Pre-infusion Anti-OBI-1 Antibody Titers, the Total Dose of OBI-1, the Outcome at 24 Hours and the Eventual Control of the Bleeding Episode
Time Frame: Through 90 days ± 7 days following final OBI-1 dose
Population: Because of expected sparseness of positive anti-OBI-1 antibody titers, formal statistical analyses of correlation were not performed.
Arm/Group | OBI-1
Number analyzed (Participants) | 0

12. Secondary Outcome: Pharmacokinetics (PK) Analysis- Plasma Clearance
Description: Participation in the PK sampling was optional. PK parameters obtained from the non-bleeding state were summarized with descriptive statistics.
Time Frame: Pre-infusion 15-20 minutes, Post-infusion 1, 3, 6, 12, 18, 24 hours
Population: PK population (= all subjects in the ITT population who consent to PK draws and have factor VIII levels measured at the central reference laboratory)
Measure: Mean (Standard Deviation); unit: U/(percent activity*hours)
Arm/Group | OBI-1
Number analyzed (Participants) | 5
U/(percent activity*hours)
  Chromogenic FVIII activity assay | 11.80 (13.44)
  One-stage FVIII activity assay | 18.07 (21.78)

13. Secondary Outcome: PK Analysis- Volume of Distribution (Vd) at Steady State
Description: as for outcome 12
Time Frame: Pre-infusion 15-20 minutes, Post-infusion 1, 3, 6, 12, 18, 24 hours
Population: PK population
Measure: Mean (Standard Deviation); unit: U/percent activity
Arm/Group | OBI-1
Number analyzed (Participants) | 5
U/percent activity
  Chromogenic FVIII activity assay | 53.8 (52.9)
  One-stage FVIII activity assay | 65.1 (45.1)

14. Secondary Outcome: PK Analysis- Area Under the Concentration-time Curve (AUC) From Time 0 to the Last Measurable Concentration
Description: Participation in the PK sampling was optional. PK parameters obtained from the non-bleeding state were summarized with descriptive statistics. AUC was calculated as area under the percent activity-time curve.
Time Frame: Pre-infusion 15-20 minutes, Post-infusion 1, 3, 6, 12, 18, 24 hours
Population: PK population
Measure: Mean (Standard Deviation); unit: percent activity*hours
Arm/Group | OBI-1
Number analyzed (Participants) | 5
percent activity*hours
  Chromogenic FVIII activity assay | 599 (459)
  One-stage FVIII activity assay | 423 (340)

15. Secondary Outcome: PK Analysis- Terminal Half-life
Description: Participation in the PK sampling was optional. PK parameters obtained from the non-bleeding state were summarized with descriptive statistics. Half-life was calculated as the time it took to reduce percent activity by half.
Time Frame: Pre-infusion 15-20 minutes, Post-infusion 1, 3, 6, 12, 18, 24 hours
Population: PK population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | OBI-1
Number analyzed (Participants) | 5
hours
  Chromogenic FVIII activity assay | 3.3 (0.4)
  One-stage FVIII activity assay | 3.5 (1.0)

16. Secondary Outcome: Number of Participants Who Developed de Novo Anti-OBI-1 Antibody Titers
Time Frame: Through 90 days ± 7 days following final OBI-1 dose
Population: 28 eligible subjects with acquired hemophilia A in the ITT population (n=29), of whom 18 had no detectable anti-porcine FVIII inhibitor titers at baseline (<0.6 BU) and 10 had detectable anti-porcine FVIII antibody titers at baseline (>=0.6 BU)
Measure: Number; unit: participants
Arm/Group | OBI-1
Number analyzed (Participants) | 28
participants | 5

17. Secondary Outcome: Number of Participants Who Developed an Anti-host Cell Protein Baby Hamster Kidney (BHK) Antibody Titer
Time Frame: Through 90 days ± 7 days following final OBI-1 dose
Population: 21 subjects in the ITT population (n=29) with available baseline and follow-up test results
Measure: Number; unit: participants
Arm/Group | OBI-1
Number analyzed (Participants) | 21
participants | 0

18. Other Pre Specified Outcome: Anti-human Factor VIII Antibody Titer
Time Frame: Through 90 days ± 7 days following final OBI-1 dose
Population: Anti-human factor VIII antibody titer data were presented in subject data listings. No statistical test was planned for anti-human factor VIII antibody titer.
Arm/Group | OBI-1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Through 90 days ± 7 days following final OBI-1 dose
Description: Subjects were monitored for adverse events from the time the subject presented with the initial bleeding episode until the end of the follow-up period.
Arm/Group | OBI-1
Serious Adverse Events (participants affected / at risk) | 13/29
Other Adverse Events (participants affected / at risk) | 27/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OBI-1 (N=29)
Asthenia (General disorders) | 1 (1) — Generalized weakness
Dizziness (Nervous system disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 2 (2)
Brain edema (Nervous system disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 2 (2)
Transient ischemic attack (Nervous system disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Systemic mycosis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (2)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Hemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Intestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OBI-1 (N=29)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 12 (12)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Mouth ulceration (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (5)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Peripheral edema (General disorders) | 6 (7)
Pyrexia (General disorders) | 3 (5)
Bacteremia (Infections and infestations) | 2 (2)
Bacteriuria (Infections and infestations) | 2 (2)
Candidiasis (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 3 (3)
Oral candidiasis (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2)
Antibody test positive (Investigations) | 2 (2) — Positive OBI-1 (anti-porcine FVIII) inhibitor test result
Troponin I increased (Investigations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 7 (11)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Muscle hemorrhage (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 3 (4)
Hypotension (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Due to the low number of subjects available for evaluation, statistical tests could only be performed for the primary outcome measure. The results of all other outcome measures are descriptive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For this study, PIs are restricted from independently publishing results before completion of a single multicenter publication or one year after study completion, whichever occurs first. Baxter requires a review of results communications (eg, for confidential information) ≥30 days prior to submission or communication. Baxter may request an additional delay of ≤60 days (eg, if a patentable invention is disclosed).